CLINICAL TRIAL: NCT00997646
Title: Performance of a Hospitalist-run Ward: a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chin-Chung Shu, National Taiwan University Hospital
Other Study IDs: 200910008R
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Performance of a Hospitalist-run Ward
Keywords: Performance; hospitalist; ward; hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients in hospitalist-run ward: Patients was admitted from ER to a hospitalist-run ward.
- Patients in conventional ward: Patients was admitted from ER to a non hospitalist-run ward.

SUMMARY:
To realize performance of a new system - hospitalist-run ward in Taiwan.

DETAILED DESCRIPTION:
The emergency department (ED) of National Taiwan University hospital manages a large amount of patients load in Taipei metropolitan. The short-stay unit in our ED is a pool for those needing observation or following management. However, the length of ED stay seems to be longer than those reported in western literature. It might be caused by limited facility availability of our ward. Actually, the bed vacancy of our ward is not only reserved for patients from ED but also for those from outpatients or other hospitals. A full ward for taking over the patients from ED only might be a solution in the future. However, internists and surgeons who care most of hospitalized patients are currently believed not a career priority because of their high risk and loading but relative low payment by National Health insurance in Taiwan. Under the deficiency of residents for patient-care, a system of hospitalist-run ward should be established.

The role of hospitalist, an in-patient physician, has been discussed since 1996. The pros and cons were debated controversially. The disadvantage is that the continuity of patient care will be interrupted by primary care physician. In addition, discharged summary are usually not completed in following clinic. On the other hand, the hospitalists need less cost than internists in recent studies but the quality and safety was considered similar. Actually, it is widely accepted that hospitalist can do an efficient job of handling inpatient admissions. The field has also continued to grow worldwide in recent decades. A hospitalist-run ward becomes more frequent for common but relatively low risk diseases including exacerbation of chronic obstructive pulmonary disease, pneumonia, urinary tract infection, ischemic stoke, cellulitis and congestive heart failure. Of course, some disease entities need longer length of hospital stay in nature.

We are thus interested in the efficiency of a hospitalist-run ward in Taiwan. Therefore, we set up a hospitalist-run ward for taking over the patients who needed hospitalization from our ED and observe the performance of the ward and the outcome of the in-patients.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* admitted from Emergency department

Exclusion Criteria:

* without informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who was admitted to a hospitalist-run ward
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Cost and quality of this hospitalization | 2 years

SECONDARY OUTCOMES:
Mortality and morbidity of this hospitalization | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan